CLINICAL TRIAL: NCT06950229
Title: Efficacy and Safety of Povidone Iodine Versus Normal Saline in Preoperative Vaginal Cleansing Before Caesarean Section: A Randomized Controlled Trial
Brief Title: Povidone Iodine Versus Normal Saline in Preoperative Vaginal Cleansing Before Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Teaching Hospital Abakaliki (Other Government)
Responsible Party: Principal Investigator, Assumpta Nnenna Nweke, Principal Investigator, Federal Teaching Hospital Abakaliki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AE-FUTHA/REC/VOL3/2020/069
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Povidone Iodine; Normal Saline; Pre-operative
Keywords: Povidone Iodine; Normal Saline; Caesarean section; vaginal cleansing
MeSH Terms: interventions — Povidone-Iodine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Povidone group (Active Comparator): Hundred (100) ml of 5% povidone iodine was poured into a sterilized bowl (galipot). Three pieces of gauze held with sponge holding forceps was dipped into the sterilized bowl containing 100mls of 5% povidone iodine and was allowed to be well soaked with 5% povidone iodine and thereafter used to swab the vulva in 360 degrees. one gram of ceftriaxone and 500mg of metronidazole was given prior to the procedure.
  Interventions: Drug: Povidone-Iodine
- Normal Saline (Experimental): Hundred (100) ml of Normal saline was poured into a sterilized bowl (galipot). Three pieces of gauze held with sponge holding forceps was dipped into the sterilized bowl containing 100mls of Normal saline and was allowed to be well soaked with Normal saline and thereafter used to swab the vulva in 360 degrees. one gram of ceftriaxone and 500mg of metronidazole was given prior to the procedure.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Povidone-Iodine — Hundred (100) ml of 5% povidone iodine was poured into a sterilized bowl (galipot). Three pieces of gauze held with sponge holding forceps was dipped into the sterilized bowl containing 100mls of 5% povidone iodine and was allowed to be well soaked with 5% povidone iodine and thereafter used to swab the vulva in 360 degrees. one gram of ceftriaxone and 500mg of metronidazole was given prior to the procedure.
  Arms: Povidone group
Drug: Normal Saline — Hundred (100) ml of Normal saline was poured into a sterilized bowl (galipot). Three pieces of gauze held with sponge holding forceps was dipped into the sterilized bowl containing 100mls of Normal Saline and was allowed to be well soaked with Normal saline and thereafter used to swab the vulva in 360 degrees. one gram of ceftriaxone and 500 mg of metronidazole was given prior to the procedure.
  Arms: Normal Saline

SUMMARY:
Post-caesarean maternal infectious morbidity is still a big challenge despite prophylactic antibiotics and preoperative vaginal cleansing with povidone-iodine use in reduction of post-caesarean endometritis.Povidone iodine has been found to cause significant irritation to the vaginal mucosa especially in females with iodine hypersensitivity necessitating the study of efficacy of normal saline which has minimal side effects in the prevention of post caesarean complications

DETAILED DESCRIPTION:
BACKGROUND: Maternal infectious morbidity is a common complication of caesarean section and is the third leading cause of maternal mortality in Nigeria and account for 15% of maternal death worldwide. Post-caesarean maternal infectious morbidity is still a big challenge despite prophylactic antibiotics and other modalities adopted to prevent it. Recently, preoperative vaginal cleansing with povidone-iodine (PI) was recommended in reduction of post-caesarean endometritis, but this may lead to significant irritation to the vaginal mucosa resulting from allergic reactions in females with iodine hypersensitivity. Normal saline (NS) is an effective cleaning solution and doesn't have allergic effect on healthy tissues. It is accessible, non-irritant, and less expensive in contrast to povidone iodine.

AIM: To compare the difference in the incidence of postoperative vaginal irritation symptoms and the rate of postoperative infections after using Povidone iodine versus Normal saline solution in vaginal cleansing before caesarean section at the Alex Ekwueme Federal University Teaching Hospital Abakaliki.

METHODOLOGY: This was a randomized controlled trial involving two hundred and twenty four (224) consenting pregnant women undergoing caesarean section in AE-FUTHA. These women were grouped into two arms; group 1 (Vaginal cleansing with povidone iodine) and group 2 (vaginal cleansing with normal saline solution). Both groups received prophylactic antibiotics and anterior abdominal wall scrubbing. Subsequently, the researcher and assistant reviewed the patients for infectious

morbidity daily during ward rounds till discharge and vaginal irritation symptoms 24hours postoperatively, and daily during ward round till discharge.

DATA ANALYSIS: Data was analyzed using statistical Package for Social Science (IBM SPSS) software (version 20, Chicago II, USA). Continuous variables were presented as mean and standard deviation (Mean ± SD), while categorical variables were presented as numbers, frequencies and percentages. Student t- test (t-test) was used for comparison between groups for quantitative variables while the chi- square was performed for comparing categorical variables. Relative risk and 95% confidence interval were calculated for outcome measures. A difference with a P value of < 0.05 was taken to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

. All consenting parturient for either elective or emergency caesarean section after the age of viability

Exclusion Criteria:

* Women with known allergy to topical povidone-iodine.
* Women with presence of pre-existing vaginal irritation symptoms as itching, burning, swelling and vaginal pain.
* Antepartum haemorrhage (Placenta praevia).
* Cord prolapse
* Clinical evidence of Chorioamnionitis
* Face presentation with ruptured membranes to avoid contact of fetal face with iodine.
* Women with immunosupression due to HIV/AIDS, Diabetes Miletus or chronic use of steroids.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 224 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Post caesarean endometritis. | 24 hours
  Patient that has at least two or more of the following signs and symptoms with no other recognized cause: fever greater than or equal to 380c, abdominal pain, uterine tenderness and purulent drainage from the uterus
Post operative vaginal irritation | 24 hours
  presence of symptoms like itching, burning, swelling and vaginal pain following the vaginal cleansing with either 5% povidone iodine or normal saline solution.

CONTACTS AND LOCATIONS:
Locations (1):
- Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No